CLINICAL TRIAL: NCT05224427
Title: A Pilot Study of Reducing Test-Anxiety in a Cohort of Underrepresented in Medicine MCAT Students Using Near-Peer Coaching
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: PRO00035403
Record Dates: First submitted 2022-01-25; First posted 2022-02-04 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Test Anxiety

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Near-Peer Coaching — Targeted coaching by near-peer medical students

SUMMARY:
We elected to establish a pilot near-peer coaching program for URM students enrolled at the Medical College of Wisconsin MCAT program. We quantified baseline and specific time point test-anxieties using the validated Westside test anxiety scale. We asked about MCAT concerns and program impressions via a free response section and analyzed results with inductive analysis.

DETAILED DESCRIPTION:
The proposed study occurred in-person at the Medical College of Wisconsin or online via video conferencing. The proposed study designs were approved by the Institution's Review Board (PRO00035403). A previous Medical College of Wisconsin ( MCW) MCAT-training program for URM students was started in 2017 and enrolled all twenty-two students from this program within the first year, and all twelve students the second year. All participants enrolled in the MCAT program were from Wisconsin and attended undergraduate or finished undergraduate studies within the past 5 years and were intending to apply to medical school.

Volunteer near-peer mentors were recruited from existing MD or MD PhD candidates at MCW. Coaches were oriented at the beginning of each program year, and periodically sent reminders and instructions on what to cover. Initial MCAT coaching meetings were instructed to cover study schedules, effective studying and exam strategy while later coaching meetings recommended coaches share their stories of how they dealt with test-anxiety, strategies to deal with test-anxiety (i.e. visit the test-center a week before , positive mentality about wrong answers during practice, and increasingly practicing under test-day conditions), and for open discussion with the student about how they were feeling. In response to student concerns about feeling limited by these topics, coaches were no longer instructed, rather recommended these topics to be covered in the second year of the program.

Students were consented and oriented in a group or individual setting and surveys were distributed via QualtricsXM for baseline, after a mock MCAT exam four months before most exam dates, and after each MCAT Coaching meeting. In the first year of the program between 2019-2020, three official MCAT coaching sessions were scheduled: one every three months starting in August. In response to student concerns, the second year of the program continued with the three official MCAT coaching sessions, while explicitly stating that students can meet as many times as they wish above this number. Due to COVID-19, an in-person mock MCAT time point was not possible in the second iteration.

Surveys were anonymous and tracked using a pin. Surveys measured quantitative test-anxiety scores using the validated Westside test-anxiety scale. The mean and the standard deviation were calculated in excel. Significance was calculated first using an F-test to determine the variances between the populations, followed by using the appropriate two-tailed student's t-test in Excel. Statistical significance was p<0.05. Qualitative data regarding student concerns regarding the MCAT as well as comments on the program were elicited via free response. A sample of the survey is available in Figure 1. Inductive analysis was performed on the free response answers. They were categorized into various themes using line-by-line coding. Sentences within the answers could overlap into different themes or not be related to any theme.

ELIGIBILITY:
Inclusion Criteria:

* From Wisconsin
* Attended undergraduate or finished undergraduate studies within the past 5 years and were intending to apply to medical school.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All participants were enrolled in a previous Medical College of Wisconsin ( MCW) MCAT-training program for URM students was started in 2017, were also from Wisconsin and attended undergraduate or finished undergraduate studies within the past 5 years and were intending to apply to medical school.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Test-anxiety as measured by the West-side test anxiety scale | 1 year

SECONDARY OUTCOMES:
Qualitative MCAT concerns | 1 year
Qualitative feedback about coaching | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liu, B., Hodge, A., Jushka, C., & Hueston, W. J. (2022). A Pilot Study of Reducing Test Anxiety in a Cohort of Underrepresented in Medicine MCAT Students Using Near-Peer Coaching. International Journal of Medical Students, 10(2), 139-147. https://doi.org/10.5195/ijms.2022.1185 (Original work published June 30, 2022)